CLINICAL TRIAL: NCT03911518
Title: Loop vs. Traditional Incision and Drainage: A Randomized Controlled Pilot Trial
Brief Title: Loop Drainage Versus Incision and Drainage for Abscesses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot study not necessary as new data has become available.
Sponsor: Gary Peksa (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other); Loyola University (Other); Kaiser Permanente (Other); Stony Brook University (Other)
Responsible Party: Sponsor-Investigator, Gary Peksa, Co-investigator; Assistant Professor, Emergency Medicine, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19021803
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Abscess of Skin and/or Subcutaneous Tissue
Keywords: incision and drainage; loop drainage; soft tissue infection; abscess
MeSH Terms: conditions — Surgical Wound; Soft Tissue Infections; Abscess | interventions — Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An investigator blinded to treatment assignment determine the cosmetic healing rate at 90 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Incision and drainage.
  Interventions: Procedure: Incision and drainage
- Intervention (Experimental): Loop drainage.
  Interventions: Procedure: Loop drainage

INTERVENTIONS:
Procedure: Loop drainage — Loop drainage will occur via 2 small incisions, approximately 2 cm, with the cuff from the base of a sterile glove pulled through and then tied off.
  Arms: Intervention
Procedure: Incision and drainage — The wound will be incised with a #11 blade scalpel along the point of maximal fluctuance, approximately 2-3 cm, and then all loculations bluntly dissected with a set of Kelly clamps. After drainage of pus, the wound will be loosely packed with gauze.
  Arms: Control

SUMMARY:
This is a multicenter randomized controlled trial of loop drainage versus traditional incision and drainage in adult patients presenting to the emergency department.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

The usual care in the United States for abscess management is generally incision and drainage. There have been various techniques described for incision and drainage: 1. incision and drainage followed by healing by secondary intention, 2. Incision and drainage followed by primary closure, and 3. Loop drainage (more recently, the topic of this study) with subsequent loop removal and healing by secondary intention. The treatment failure rate for traditional incision and drainage is variable, but can range from 10-30%. Costs associated with treatment failure are between $1,000 and $2,0005. The relatively high failure rate associated with traditional incision and drainage has led to research into less invasive, more effective techniques. In 2010, the loop drainage technique was first described. This technique consists of making 2 small incisions on either end of the abscess cavity followed by pulling a small drain through the incisions and then tying the drain in place. It remains in place and is removed once no further drainage is noticed (usually in 10-14 days). Original studies were primarily done by pediatric surgeons using vessel loops or penrose drains.

In 2014, the concept of using the cuff from the bottom of a sterile glove was introduced. This allows for this technique to easily be used with materials found easily in any emergency department. The amount of research done with this technique on adults is limited. To date, only two studies with a total of 109 patients evaluated loop drainage in adults. One of these studies was retrospective and included only 63 patients. The other prospective study was limited in that it included only 46 patients. Given the demonstration of increased clinical cure rate in pediatric populations and the potential for increased clinical cure rates in adults, more study into this topic is worthwhile to determine the optimal approach to adult subcutaneous abscess drainage.

STUDY DESCRIPTION

This study will be a pilot study and multi-center prospective randomized controlled trial evaluating loop drainage compared to conventional incision and drainage in adults older than 18 who have simple, purulent, cutaneous abscesses deemed amenable to outpatient incision and drainage by the attending clinician.

Study participants will be randomized to investigational vs control arm in a 1:1 ratio (Randomization will occur via blocked randomization in blocks of 10). Enrollment will occur primarily when investigators are on shift (convenience sampling). This study will not be blinded, however, observer bias will be reduced by having an investigator blinded to treatment assignment determine the cosmetic healing rate at 90 days.

Participants will receive drainage of their abscess (either conventional or loop). For conventional drainage, the wound will be incised with a #11 blade scalpel along the point of maximal fluctuance, approximately 2-3 cm, and then all loculations bluntly dissected with a set of Kelly clamps. After drainage of pus, the wound will be loosely packed with gauze. Afterwards, a dry dressing will be placed and the patient will be instructed to change the external dressing twice daily or every time it becomes saturated. Patients randomized to standard care will be instructed to remove the packing at 48 hours after incision and drainage.

Loop drainage will occur via 2 small incisions, approximately 2 cm, with the cuff from the base of a sterile glove pulled through and then tied off3. The patient will be instructed to move this cuff back and forth three times daily and cover it with a dry dressing.

Once the abscess drainage procedure is complete, the participant will complete a questionnaire asking about pain during procedure and satisfaction with the procedure. All participants will be discharged with a prescription trimethoprim-sulfamethoxazole (TMP-SMX) 160mg/800mg, two tablets by mouth twice daily for ten days. All participants will be instructed to return to the emergency department and contact the PI if they have any worsening signs of infection. Between 10 and 14 days after the initial procedure, patients will follow up in the emergency department for wound recheck. At this visit, the maximal diameter of both erythema and swelling will be measured, and a questionnaire will be administered regarding wound care satisfaction, repeat medical visits, fevers, and any side effects of either the procedure or antibiotic therapy. Loop participants will have the loop removed at the follow up visit. Participants will be called at 30 days for data collection on abscess recurrences. Patient will be asked to return for a wound recheck and submit a photo of the wound, to assess cosmetic appearance of wound at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Abscess is considered simple, purulent, and cutaneous
* Abscess is deemed amenable to outpatient drainage

Exclusion Criteria:

* Inability to speak English
* Abscess location of breast or face
* Pilonidal abscesses
* Concurrent use of chemotherapy or steroids
* Allergy to sulfa/trimethoprim or lidocaine
* Inability to provide consent
* Incarcerated patients
* Inability to give a valid contact number or email address
* Presence of multiple abscesses
* Abscess size less than 2 cm
* Pregnant patients
* History of glucose-6-phosphate dehydrogenase deficiency
* History of Steven Johnson's Syndrome
* Patients with fever greater than 100.4 Fahrenheit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical Cure | Days 10-14
  Defined as healing of the abscess without the need for further clinical intervention (change in antibiotics, repeat drainage, or admission)

SECONDARY OUTCOMES:
Intra-Procedure Pain Rating | Day 0
  Numeric rating scale of 0-10. A rating of 0 indicates no pain. A rating of 10 indicates the worst pain.
Time to Complete Drainage | Day 0
  Time from initial incision to application of dry dressing
Patient Satisfaction: Numeric rating scale | Days 0, 10-14
  Likert scale of 1-5. A rating of 1 indicates poor satisfaction. A rating of 5 indicates the best satisfaction.
Provider Satisfaction: Numeric rating scale | Day 0
  Likert scale of 1-5. A rating of 1 indicates poor satisfaction. A rating of 5 indicates the best satisfaction.
Recurrence Rate | Day 30
  New lesions requiring drainage
Cosmetic Healing | Day 90
  Visual analog scale of 1-100 mm. A score of 1 indicates poor cosmetic healing. A score of 100 indicates excellent cosmetic healing.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Schmitz, MD, Principal Investigator — Uniformed Services University of the Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ladde JG, Baker S, Rodgers CN, Papa L. The LOOP technique: a novel incision and drainage technique in the treatment of skin abscesses in a pediatric ED. Am J Emerg Med. 2015 Feb;33(2):271-6. doi: 10.1016/j.ajem.2014.10.014. Epub 2014 Oct 16. PMID 25435407
- [Background] Thompson DO. Loop drainage of cutaneous abscesses using a modified sterile glove: a promising technique. J Emerg Med. 2014 Aug;47(2):188-91. doi: 10.1016/j.jemermed.2014.04.035. Epub 2014 Jun 11. PMID 24928539
- [Background] Stevens DL, Bisno AL, Chambers HF, Dellinger EP, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan SL, Montoya JG, Wade JC; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of skin and soft tissue infections: 2014 update by the Infectious Diseases Society of America. Clin Infect Dis. 2014 Jul 15;59(2):e10-52. doi: 10.1093/cid/ciu444. PMID 24973422
- [Background] McNamara WF, Hartin CW Jr, Escobar MA, Yamout SZ, Lau ST, Lee YH. An alternative to open incision and drainage for community-acquired soft tissue abscesses in children. J Pediatr Surg. 2011 Mar;46(3):502-6. doi: 10.1016/j.jpedsurg.2010.08.019. PMID 21376200
- [Background] Gaszynski R, Punch G, Verschuer K. Loop and drain technique for subcutaneous abscess: a safe minimally invasive procedure in an adult population. ANZ J Surg. 2018 Jan;88(1-2):87-90. doi: 10.1111/ans.13709. Epub 2016 Sep 12. PMID 27621209
- [Background] Ozturan IU, Dogan NO, Karakayali O, Ozbek AE, Yilmaz S, Pekdemir M, Suner S. Comparison of loop and primary incision & drainage techniques in adult patients with cutaneous abscess: A preliminary, randomized clinical trial. Am J Emerg Med. 2017 Jun;35(6):830-834. doi: 10.1016/j.ajem.2017.01.036. Epub 2017 Jan 22. PMID 28162873
- [Background] Gottlieb M, Peksa GD. Comparison of the loop technique with incision and drainage for soft tissue abscesses: A systematic review and meta-analysis. Am J Emerg Med. 2018 Jan;36(1):128-133. doi: 10.1016/j.ajem.2017.09.007. Epub 2017 Sep 10. PMID 28917436